CLINICAL TRIAL: NCT04477122
Title: Effects of Radial Shock Wave Therapy in the Treatment of Temporomandibular Joint Syndrome. A Randomized Clinical Trial
Brief Title: Effects of Radial Shock Wave Therapy in the Treatment of Temporomandibular Joint Syndrome.
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Jaén (Other)
Responsible Party: Principal Investigator, Alfonso Javier Ibáñez-Vera, Health Sciences Department Professor, University of Jaén
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: UJaen Posture
Record Dates: First submitted 2020-07-07; First posted 2020-07-20 (Actual); Last update posted 2021-01-29 (Actual); Status verified 2021-01

CONDITIONS: Temporomandibular Joint Disorders; Temporomandibular Joint Dysfunction Syndrome
Keywords: temporomandibular joint; temporomandibular joint syndrome; temporomandibular joint dysfunction; extracorporeal shock waves
MeSH Terms: conditions — Temporomandibular Joint Disorders; Temporomandibular Joint Dysfunction Syndrome | interventions — Musculoskeletal Manipulations

STUDY DESIGN:
Intervention Model Description: Two groups: experimental one and placebo group, receiving the intervention at the same time
Who Masked: Participant, Investigator, Outcomes Assessor
Masking Description: Participants will take and opaque enveloped who revealed the allocation group (named as RED or BLUE for blindness conditions). Investigators will not be aware of the which device is sham or real treatment due to codification. The outcomes assessor will be a different person from the investigator and the care providers, unaware of group allocation and treatment.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Blue (Experimental): Four sessions (one per week along one month) of manual therapy (25 minutes of massage on temporal, masseter and pterygoid muscles and 5 minutes of joint passive mobilization) and 3 minutes (2000 shots approximately) of extracorporeal radial shock waves therapy on painful points of masseter and temporal muscles at 2 bars and 10 Hertzs. Participants will wear splint 23 hours/day
  Interventions: Other: Manual therapy and extracorporeal radial shock waves therapy
- Red (Placebo Comparator): Four sessions (one per week along one month) of manual therapy (25 minutes of massage on temporal, masseter and pterygoid muscles and 5 minutes of joint passive mobilization) and 3 minutes of placebo extracorporeal radial shock waves therapy on painful points of masseter and temporal muscles. Participants will wear splint 23 hours/day
  Interventions: Other: Manual therapy and extracorporeal radial shock waves therapy

INTERVENTIONS:
Other: Manual therapy and extracorporeal radial shock waves therapy — 25 minutes of manual therapy, 5 minutes of temporomandibular joint mobilization and 3 minutes of extracorporeal radial shock waves therapy (real or placebo)

SUMMARY:
The aim of this study is to assess the effects of radial shock wave therapy in the treatment of temporomandibular joint syndrome. For this objective, subjects recruited will be allocated in an experimental group or a placebo group. Both groups will receive one manual therapy and radial shock waves therapy (real for experimental group, a sham device for placebo group) session per week along one month. Pain, neck function and quality of life measured will be performed before the intervention, after the last treatment and at one month follow-up.

DETAILED DESCRIPTION:
Temporomandibular Disorders (TMDs) are a subgroup of painful orofacial disorders of the stomatognathic system, characterized by TemporoMandibular Joint (TMJ) pain, fatigue of the cranio-cervico-facial muscles (especially the masticatory muscles), limitation of mandibular movement and the presence of a click or crackling sound in the ATM.

The main signs and symptoms associated with TMDs are bruxism (33%), myofascial pain (14%), headache (96%) and functional limitation (93%), the latter being related to posture.

The quality of life of patients with TMD involvement is diminished in various facets of their lives, leading to a private expense for the patient as well as a public expense resulting from a poor referral due to the lack of adequate treatment for TMDs. This expense ranges in Spanish public hospitals at € 146.9 with a minimum of € 52 and a maximum of € 425.

From this study, we are going to carry out a non-invasive, analgesic, anti-inflammatory treatment and without negative side effects for the patient through radial extracorporeal shock waves (rESWT), and manual therapy (TM).

Among the effects produced by shock waves we find that they improve circulation due to increased blood flow and oxygenation, at tissue level the permeability of the membrane increases and its metabolic process, therefore facilitating the activation of tissue regeneration processes experiencing dystrophic changes. Furthermore, shock waves cause anti-inflammatory effects and muscle relaxation.

The main objective of the study is to evaluate the capacity of the shock waves to improve the alterations due to temporomandibular disorders. To meet the above objective, a single-blind randomized clinical trial study has been designed. The selected subjects will be of legal age diagnosed with temporomandibular disorder and those subjects that due to their own characteristics are not able to carry out the study will be excluded. Subjects will receive a weekly physical therapy session for four weeks. Subjects will be randomly assigned to two groups: T1 intervention group consisting of subjects who will receive manual therapy treatment and shock waves and T2 placebo group in which the subjects will receive manual therapy and placebo shock waves.

Subjects will be evaluated using sociodemographic variables such as age, sex, weight, height, Body Mass Index, educational level, work, smoking, alcohol and physical activity and function tests and quality of life questionnaires will be used. Measurements will be made pre and post-treatment, one month after the last evaluation, the measurements will be made again for follow-up. The intervention will be one day a week for four consecutive weeks.

The data will be collected using a self-implementing questionnaire, these data will be transferred to an excel table and then transferred to SPSS 19.0 (SPSS Inc., Chicago, IL) and MedCalc 19.1 (MedCalc Software Bv, Ostend, Belgium, http: // wwww .medcalc.org; 2019) for the subsequent statistical analysis, the data being stripped of any direct reference to the subject to preserve confidentiality.

The descriptive analysis will be carried out with means and standard deviations for continuous variables, frequencies and percentages for categorical variables. The normality of the continuous variables will be calculated with the Kolmogorov-Smirnov test and the homocedasticity of the sample with the Levene test.

All the statistical analysis will be carried out with a confidence level of 95% (p <0.05), for the comparison of the two groups we will use the Student's t-test and the Chi-square test. Comparisons between treatment group and placebo group will be made using repeated measures analysis of variance and ANOVA, followed by Bonferroni to compare measures replicated over time.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosed of temporomandibular disorder by medical doctor.

Exclusion Criteria:

* Subjects who due to their own characteristics are not able to carry out the study tests

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 63 (Actual)
Dates: Start 2020-10-27 (Actual); Primary Completion 2020-12-29 (Actual); Study Completion 2021-01-25 (Actual)

PRIMARY OUTCOMES:
Temporomandibular joint pain | Baseline
  Actual local pain at temporomandibular joint measured with Numerical pain rating scale
Temporomandibular joint pain | At one month
  Actual local pain at temporomandibular joint measured with Numerical pain rating scale
Temporomandibular joint pain Temporomandibular joint pain | At two months
  Actual local pain at temporomandibular joint measured with Numerical pain rating scale
Neck function | Baseline
  Neck Disability Index, a 10 questions scale about neck function
Neck function | At one month
  Neck Disability Index, a 10 questions scale about neck function
Neck function | At two months
  Neck Disability Index, a 10 questions scale about neck function

SECONDARY OUTCOMES:
Pain threshold | Baseline
  Beginning of pain feeling referred at pressure with algometer at temporomandibular joint
Pain threshold | At one month
  Beginning of pain feeling referred at pressure with algometer at temporomandibular joint
Pain threshold | At two months
  Beginning of pain feeling referred at pressure with algometer at temporomandibular joint
Headache impact in quality of life | Baseline
  Headache Impact Test (HIT-6) consisting on six questions
Headache impact in quality of life | At one month
  Headache Impact Test (HIT-6) consisting on six questions
Headache impact in quality of life | At two months
  Headache Impact Test (HIT-6) consisting on six questions
Dizziness | Baseline
  Dizziness measured with Dizziness Handicap Inventory, 25 questions about the impact of dizziness in patient's life
Dizziness | At one month
  Dizziness measured with Dizziness Handicap Inventory, 25 questions about the impact of dizziness in patient's life
Dizziness | At two months
  Dizziness measured with Dizziness Handicap Inventory, 25 questions about the impact of dizziness in patient's life
Quality of life Measured with SF-12 | Baseline
  12 questions about quality of life perceived
Quality of life Measured with SF-12 | At one month
  12 questions about quality of life perceived
Quality of life Measured with SF-12 | At two months
  12 questions about quality of life perceived
Temporomandibular joint function | Baseline
  Fonseca Anamnesis Index, 10 questions about temporomandibular joint function
Temporomandibular joint function | At one month
  Fonseca Anamnesis Index, 10 questions about temporomandibular joint function
Temporomandibular joint function | At two months
  Fonseca Anamnesis Index, 10 questions about temporomandibular joint function
Temporomandibular joint function | Baseline
  Short form of Fonseca Anamnesis Index, 5 questions about temporomandibular joint function
Temporomandibular joint function | At one month
  Short form of Fonseca Anamnesis Index, 5 questions about temporomandibular joint function
Temporomandibular joint function | At two months
  Short form of Fonseca Anamnesis Index, 5 questions about temporomandibular joint function

CONTACTS AND LOCATIONS:
Locations (1):
- Clinica Fisiomedic, Seville, Spain

IPD SHARING:
Plan to Share IPD: No
Data will be available under request to the authors/promotor